CLINICAL TRIAL: NCT04988100
Title: Impact of Splenic Artery Ligation in Living Donor Liver Transplantation for Patients With Portal Hypertension on Early Graft Function.
Brief Title: Impact of Splenic Artery Ligation in LDLT for Patients With Portal Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Rashad Abdelaziz, Principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIM in LDLT
Record Dates: First submitted 2021-07-25; First posted 2021-08-03 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Living Donor Liver Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who undergo Splenic artery ligation (Experimental): If inclusion criteria are met, these group of patients will undergo splenic artery ligation .
  Interventions: Procedure: splenic artery ligation
- No splenic artery ligation (Active Comparator): If inclusion criteria are met, these group of patients will not undergo splenic artery ligation.
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: splenic artery ligation — Splenic artery will be ligated just after takeoff from coeliac trunk at the level of body of pancreas
  Arms: Patients who undergo Splenic artery ligation
Procedure: No intervention — Splenic artery is not ligated despite the presence of portal hyperperfusion
  Arms: No splenic artery ligation

SUMMARY:
In this study, the investigators aim to prove that performing splenic artery ligation in living donor liver transplantation for patients with portal hypertension is beneficial for early graft function postoperatively. The investigators will be analyzing trend of LFT's (liver function tests) after surgery, time for normalization of bilirubin, INR (international normalised ratio) and decrease in ascites, morbidity, mortality, ICU (intensive care unit) and total hospital stay.

DETAILED DESCRIPTION:
Liver transplantation (LT) is the principal treatment for end-stage liver diseases and selected cases of liver neoplasms . Living donor liver transplantation (LDLT) serves as a sole source of liver graft in some countries that do not allow donation from deceased donors for cultural, social, or religious reasons.

Hyperperfusion plays an important role in liver regeneration after LDLT, but it may induce injury in the graft . After the reperfusion of a partial graft, there is a significant increase in the portal flow, but Hepatic artery flow remains constant . Excessive portal vein flow may induce injuries in grafts and may contribute to poor graft function.

For satisfactory graft function early after LT, the portal vein pressure (PVP) value after reperfusion should be <15 mm Hg. PVP is the most important hemodynamic factor influencing the functional status of the liver and graft regeneration after LT.

The use of Splenic Artery Ligation (SAL) as a simple and safe method to modulate portal flow has been reported .

The investigators will evaluate that Splenic artery ligation in living donor liver transplantation for patients with Portal hypertension is feasible and efficient technique to improve early graft function and to decrease morbidity and hospital stay and improve outcomes .

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing Living Donor Liver Transplantation(LDLT) accepted according to hospital protocol.
* Patients who have Portal Venous Pressure (PVP) > 15 mm Hg after reperfusion .

Exclusion Criteria:

* Patients who have Portal Venous Pressure (PVP) > 15 mm Hg after reperfusion.
* Patients who had splenectomy.
* Patients who have splenic artery aneurysm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of early graft dysfunction | first postoperative month
  Number of patients who develop early graft dysfunction in each group
Time to normalisation of ascites output | first postoperative month
  time to normalisation of ascites output (in days)
Time to normalisation of INR | first postoperative month
  time to normalisation of INR (in days)
Time to normalisation of bilirubin | first postoperative month
  time to normalisation of bilirubin (in days)

SECONDARY OUTCOMES:
Morbidity | first postoperative month
  Morbidity as per Clavein Dindo classification
ICU stay | first postoperative month
  Duration of ICU stay (in days)
Mortality | first postoperative month
  death
Total hospital stay | first postoperative month
  duration of total stay in hospital after liver transplantation (in days)

REFERENCES:
- [Background] Gad EH, Alsebaey A, Lotfy M, Eltabbakh M, Sherif AA. Complications and mortality after adult to adult living donor liver transplantation: A retrospective cohort study. Ann Med Surg (Lond). 2015 Apr 25;4(2):162-71. doi: 10.1016/j.amsu.2015.04.021. eCollection 2015 Jun. PMID 26005570
- [Background] Abdeldayem H, Kashkoush S, Hegab BS, Aziz A, Shoreem H, Saleh S. Analysis of donor motivations in living donor liver transplantation. Front Surg. 2014 Jul 8;1:25. doi: 10.3389/fsurg.2014.00025. eCollection 2014. PMID 25593949
- [Background] Umeda Y, Yagi T, Sadamori H, Matsukawa H, Matsuda H, Shinoura S, Mizuno K, Yoshida R, Iwamoto T, Satoh D, Tanaka N. Effects of prophylactic splenic artery modulation on portal overperfusion and liver regeneration in small-for-size graft. Transplantation. 2008 Sep 15;86(5):673-80. doi: 10.1097/TP.0b013e318181e02d. PMID 18791439
- [Background] Ito T, Kiuchi T, Yamamoto H, Oike F, Ogura Y, Fujimoto Y, Hirohashi K, Tanaka AK. Changes in portal venous pressure in the early phase after living donor liver transplantation: pathogenesis and clinical implications. Transplantation. 2003 Apr 27;75(8):1313-7. doi: 10.1097/01.TP.0000063707.90525.10. PMID 12717222
- [Background] Jiang SM, Zhou GW, Zhang R, Peng CH, Yan JQ, Wan L, Shen C, Chen H, Li QY, Shen BY, Li HW. Role of splanchnic hemodynamics in liver regeneration after living donor liver transplantation. Liver Transpl. 2009 Sep;15(9):1043-9. doi: 10.1002/lt.21797. PMID 19718645
- [Background] Garcia-Valdecasas JC, Fuster J, Charco R, Bombuy E, Fondevila C, Ferrer J, Ayuso C, Taura P. Changes in portal vein flow after adult living-donor liver transplantation: does it influence postoperative liver function? Liver Transpl. 2003 Jun;9(6):564-9. doi: 10.1053/jlts.2003.50069. PMID 12783396
- [Result] Wu TJ, Dahiya D, Lee CS, Lee CF, Chou HS, Chan KM, Lee WC. Impact of portal venous hemodynamics on indices of liver function and graft regeneration after right lobe living donor liver transplantation. Liver Transpl. 2011 Sep;17(9):1035-45. doi: 10.1002/lt.22326. PMID 21542130